CLINICAL TRIAL: NCT03553732
Title: An Electronic Registry to Improve Adherence to Active Surveillance Monitoring Among Men With Prostate Cancer at a Safety-net Hospital: A Study Protocol
Brief Title: An Electronic Registry to Improve Adherence to Active Surveillance Monitoring at a Safety-net Hospital
Status: Terminated | Type: Observational
Why Stopped: Lack of funding
Sponsor: University of California, San Francisco (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: P30HS023558-2; P30HS023558 (NIH)
Record Dates: First submitted 2018-05-16; First posted 2018-06-12 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Prostatic Neoplasms
Keywords: active surveillance; health information technology; patient safety; adherence; ambulatory; outpatient; human factors; systems engineering; vulnerable populations; chronic disease
MeSH Terms: conditions — Prostatic Neoplasms; Chronic Disease | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Active Surveillance Patients: Patients who elect to be monitored by an Active Surveillance protocol for prostate cancer
  Interventions: Other: Registry

INTERVENTIONS:
Other: Registry — Patients who are diagnosed with prostate cancer and elect to be monitored by an Active Surveillance protocol by the Urology Clinic at Zuckerberg San Francisco General Hospital and Trauma Center will be included in this group. The intervention is the implementation of a registry, designed to replace existing but suboptimal systems for tracking patients. All Active Surveillance patients monitored by the clinic will be included.

SUMMARY:
To implement and evaluate a health information technology platform designed to support the management of patients on active surveillance for prostate cancer in an urban, publicly-funded outpatient setting.

DETAILED DESCRIPTION:
We aim to implement and evaluate a health information technology (HIT) registry at an urban, public delivery system. We will use systems engineering methodologies to design, develop, and implement the platform. The platform will be implemented in the Urology clinic that cares for patients with prostate cancer. We are conducting a prospective non-randomized pilot study that will follow men who choose active surveillance as a management strategy for prostate cancer. We aim to assess the impact of the HIT registry on patient monitoring and adherence.

The HIT platform seeks to improve the monitoring and alerting functionality of existing systems. Specifically, it replaces paper-based or ineffective computer-based systems previously used by the clinic to monitor its active surveillance patients. It will be implemented clinic-wide for all patients being monitored by an active surveillance protocol. The platform is approved for clinical use and research by the San Francisco Health Network and the University of California, San Francisco.

Research involves materials that are collected for nonresearch purposes, as well as low-risk research employing survey, interview, focus group, program evaluation, and human factors methodologies. We will solicit structured feedback from registry users designed to continuously evaluate and improve performance in a clinical area to reduce patient safety gaps. Patient medical records will be reviewed, but patients monitored on the registry will not be contacted by researchers.

Procedures are in place to monitor the registry. First, quality assurance is performed by the research team, information technology analysts in the San Francisco Health Network, as well as by the third-party software provider. This includes checking that data in the platform matches source data, such as data entered in the electronic health record. In addition, users are audited on a weekly basis. A data dictionary defining variables used in the platform exists and is updated as needed. The HIT platform users include clinicians who are responsible for monitoring patients on active surveillance for prostate cancer. Patients who are enrolled in the active surveillance program will be added to the registry by a clinician. The research team will support the clinicians in data analysis, although this will be performed with population-level, de-identified data. However, if unmediated adverse events are identified by the research team, the research team will alert the clinicians appropriately. The research team will also develop training materials and conduct training sessions to ensure that all clinicians responsible for monitoring patients on active surveillance are provided with up-to-date resources and accessible support. The HIT platform is designed to supplement, but not replace, the existing electronic health record. Data on the registry will be validated with source data and users will still engage with the source data and electronic health record as appropriate clinically and operationally.

ELIGIBILITY:
Inclusion Criteria:

* Patients who elect to be managed by Active Surveillance for prostate cancer by the Urology Clinic

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Active Surveillance for prostate cancer is recommended as an initial management strategy for men with low- to intermediate-risk prostate cancer. Eligibility criteria at our institution include diagnostic prostate-specific antigen <= 10 ng/ml, clinical stage T1 or T2, Gleason scores <= 3+4, <=33% positive cores, and <= 50% tumor in any single core. Men who do not meet these eligibility criteria by elect to be managed by Active Surveillance may also be included.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-09-29 (Actual); Study Completion 2019-09-29 (Actual)

PRIMARY OUTCOMES:
Delayed follow-up - Number of days monitoring is delayed past recommended follow-up interval, | 2 years
  measured from date monitoring (e.g. prostate-specific antigen test or biopsy) is scheduled to date monitoring occurs.
Acceptability and feasibility of intervention - Semi-structured interviews | 1 year
  Acceptability and feasibility of the intervention among clinicians will be measured using the Technology Acceptance Model (Venkatesh et al). Semi-structured interviews will be conducted to assess usefulness and ease of use.

SECONDARY OUTCOMES:
Proportion of patients lost to follow-up | 2 years
  The proportion of patients who are lost to follow-up, defined as three subsequent unsuccessful outreach attempts
Proportion of patients that adhere to recommended monitoring | 2 years
  Adherence to monitoring (e.g. prostate-specific antigen test every 3 months) will be assessed. Monitoring will be considered adherent if it occurs within 30 days of the recommendation.
Proportion of patients that move from active surveillance to active treatment at a cancer stage that is more advanced than the stage recorded upon entry into program. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Urmimala Sarkar, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital and Trauma Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Venkatesh, Viswanath; Morris, Michael G.; Davis, Gordon B.; and Davis, Fred D.. 2003.
- [Derived] Cedars B, Lisker S, Borno HT, Kamal P, Breyer B, Sarkar U. An electronic registry to improve adherence to active surveillance monitoring among men with prostate cancer at a safety-net hospital: protocol for a pilot study. Pilot Feasibility Stud. 2019 Aug 14;5:101. doi: 10.1186/s40814-019-0482-x. eCollection 2019. PMID 31428442